CLINICAL TRIAL: NCT03081091
Title: Effects of Acupuncture on Pain and Quality of Life of People Affected With Chronic Widespread Pain. Study Protocol for a Randomized, Triple-blinded, Placebo Controlled Trial.
Brief Title: Effects of Acupuncture on Pain and Quality of Life of People Affected With Chronic Widespread Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat de Girona (Other)
Responsible Party: Principal Investigator, Jordi Casado Borrull, Director, Universitat de Girona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EUSESTE-CT-1
Record Dates: First submitted 2017-03-05; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Chronic Widespread Pain
MeSH Terms: conditions — Chronic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are blinded to the intervention. They will be provided with eye masks so that they cannot see which needles are used in their intervention. Moreover, the same type of equipment will be used with all the participants (although the guide tube to insert the needle is not necessary in true acupuncture).
  Given the fact that the person who carries out the intervention is different than the one assessing its effects and the latter does not know which group the evaluated subjects belong to, as well as the fact that the person responsible for the statistics is a third person who ignores which of the two groups has received true acupuncture, this is a triple-blind study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (A) Acupuncture (Active Comparator): The treatments performed will be personalized and the treatment criteria will be based on the use of the Yuan and Luo points. In clinical practice, the Yuan (source) points and the Luo (connecting) points can be used jointly, linking the two associated meridians (external-internal) in such a way that, after assessing the state of a meridian's path, its Yuan point will be combined with the Luo point of its coupled meridian and vice versa; all this depending on the condition of the muscle fibres and on the path that wants to be treated for these.
  Interventions: Device: Acupuncture
- Control group (C) Sham Acupuncture: (Sham Comparator): The course of action with the patient from the group that will use sham acupuncture will be the same as in the group that receives real treatment: patient in supine position, cleaning of the treated area, use of eye mask during the treatments and selection of points following the previously described Yuan and Luo points' criteria, based on traditional Chinese medicine.
  The difference of sham acupuncture will lie on the way of performing the acupuncture technique. It will follow the validated technique of sham acupuncture with the Park device, without needle penetration in the patient's body.
  Interventions: Device: Sham Acupuncture

INTERVENTIONS:
Device: Acupuncture — The needles used for the treatments will be single-use needles of two different gauge sizes. One size or the other will be used depending on the area to be treated and the physical condition of the patient. The needles and gauge sizes used in the study are as follows:
  Dong Bang siliconized needle 0.25 mm x 40 mm Dong Bang siliconized needle 0.20 mm x 30 mm
  The therapist will assess the patient's condition according to traditional Chinese medicine and will look at the relationship between the patient's most affected areas and the paths of the acupuncture meridians. Subsequently, the combination of Yuan and Luo points to be treated will be determined. This procedure will be followed before every acupuncture session, in such a way that the combination of the points used will depend on the evolution of the symptoms.
  Arms: Intervention group (A) Acupuncture
Device: Sham Acupuncture — It will follow the validated technique of sham acupuncture with the Park device, without needle penetration in the patient's body.
  The Park device for the performance of sham acupuncture consists of two plastic tubes, one sliding within the other, and inside which the needle created for the device slides. The longest tube is attached to a circular base, which has an adhesive surface that sticks to the skin so that the device and the needle cannot fall. Blunt ended needles will be used for this technique and thus the needle does not get to pass through the skin but produces a cutaneous stimulation similar to conventional acupuncture needles. These needles are supplied with the kit that contains the Park sham acupuncture device and are registered in the European Union as CE 0120.
  Arms: Control group (C) Sham Acupuncture:

SUMMARY:
Background: Chronic Widespread Pain (CWP) is a multidimensional disorder for which treatment as yet remains unsatisfactory. Acupuncture is one of the most sought therapeutic methods when it comes to alternative medicine, due to its minimal adverse effects and its ease of use in clinical practice. Currently, acupuncture is successfully used in China for the treatment of many chronic diseases. The work to be carried out aims to assess the effects of acupuncture on pain management and quality of life of people suffering from CWP.

Methods/design: The study is a single-center, controlled triple-blind prospective study. A total of 100 participants will be randomly distributed into two groups, the intervention group, which will receive an individualized acupuncture treatment; and control group, which will receive sham acupuncture. The treatments performed will be personalized and the treatment criteria will be based on the use of the Yuan and Luo points. They will be evaluated using a specific measurement system, constituted of the Visual Analogue Scale, The Fibromyalgia Impact Questionnaire and The Medical Outcomes Study Sleep Scale. The primary outcome measures assess whether acupuncture can bring about a decrease in pain and an improvement in the quality of life of people suffering from chronic widespread pain; the secondary outcomes assess whether the use of acupuncture leads to improved sleep quality. The results obtained will be analysed at 1st, 4th and 8th weeks from the start of treatment.

Discussion: This technique is aimed to restore some of the imbalances suffered by patients affected with CWP and to improve their symptomatology. We expect to observe a significant improvement in the pain, quality of life and sleep quality of people affected with CWP. The study will be conducted according to the STRICTA guidelines, which lay down the right way to proceed when carrying out scientific studies in the field of acupuncture.

DETAILED DESCRIPTION:
Chronic Widespread Pain (CWP) is defined as spinal pain that lasts at least three months involving both the right and left side of the body, above and below the waist.

CWP is a highly prevalent condition. According to Clauw et al., it affects 10-12% of the population and, according to Bergman et al., 10-11%. More recent studies show similar data. For their part, Mas et al. (2008) found in a nationwide study that the prevalence of fibromyalgia in Spain was of 4.2% in women and 0.2% in men, mainly in the age range between 40-49 years. All these studies have been performed in countries in the developed world and, most of the time, they have also analysed the prevalence of fibromyalgia (FM) among the same population.

Currently, acupuncture is successfully used in China for the treatment of many chronic diseases. However, in the West, the situation is quite different: acupuncture is little known and not commonly used, giving thus rise to mistrust and misunderstandings. Nevertheless, in recent years, studies have been published both in the East and in the West showing, on the one hand, the intention of traditional Chinese medicine to examine the technique and, on the other, the importance and recognition that the Western medical world is starting to bestow upon Chinese medicine.

METHODS/DESIGN

Objectives

This study seeks to meet the following objectives: assess whether acupuncture can bring about a decrease in pain and an improvement in the quality of life of people suffering from chronic widespread pain; assess whether the use of acupuncture leads to improved sleep quality.

Hypothesis

Acupuncture succeeds in reducing the pain suffered by people affected with chronic widespread pain (CWP) and in improving their quality of life. Acupuncture can improve pain and different items that have an impact on the quality of life (sleep quality and performance of daily activities).

Design

Clinical trial. Controlled triple-blind prospective study. 100 participants will be randomly distributed into two groups: intervention group (A), which will receive an individualized acupuncture treatment; and control group (S), which will receive sham acupuncture using a randomization 1:1.

Recruitment

The participants in the study will be people over 18 years old belonging to different associations of people affected with fibromyalgia from the area of Terres de l'Ebre, particularly from associations of the towns of Deltebre, Amposta, Sant Carles de la Rápita and Tortosa. Researchers will come to these entities in order to present the study in a public conference. Once the requests for participation have been received and all cases have been assessed on the basis of the inclusion and exclusion criteria, participants will be informed of the whole research process in a personal interview. After that, they will all receive an information sheet and an informed consent form, which they will be encouraged to read and sign.

Inclusion and exclusion criteria

Inclusion criteria

* Meeting the criteria set by the American College of Rheumatology for the diagnosis of chronic widespread pain.
* Accepting to sign the informed consent of participation in the study.
* Being older than 18 years.

Exclusion criteria

* Suffering from malignant diseases or active rheumatologic disorders (osteoporosis, rheumatoid arthritis, lupus erythematosus, etc.).
* Suffering from coxarthrosis or severe gonarthrosis.
* Having previously received acupuncture treatments.

Randomization

People meeting the inclusion criteria, being subsequently informed of the nature of the study and having signed the informed consent, will be assigned to one of the groups of the study. Randomization will be carried out by personnel other than the one performing the treatments and on the basis of a list obtained through the software EPIDAT (Xunta de Galicia), in such a manner that there shall be 50 people in each group: one will be treated with acupuncture according to the traditional technique to improve pain, whereas the other will act as a control group and will receive sham acupuncture. The researcher conducting the treatments will be provided with the patients' medical history together with their corresponding allocation.

Masking

Participants are blinded to the intervention. They will be provided with eye masks so that they cannot see which needles are used in their intervention. Moreover, the same type of equipment will be used with all the participants (although the guide tube to insert the needle is not necessary in true acupuncture).

Given the fact that the person who carries out the intervention is different than the one assessing its effects and the latter does not know which group the evaluated subjects belong to, as well as the fact that the person responsible for the statistics is a third person who ignores which of the two groups has received true acupuncture, this is a triple-blind study.

Intervention

The study will be conducted according to the STRICTA guidelines, which lay down the right way to proceed when carrying out scientific studies in the field of acupuncture.

Patients taking part in the trial will receive a total of 5 sessions of acupuncture (true or sham, depending on the group to which they belong within the study): 4 sessions (one per week) and a 5th session 15 days after the last one.

Intervention group (A)

The treatments performed will be personalized and the treatment criteria will be based on the use of the Yuan and Luo points. In clinical practice, the Yuan (source) points and the Luo (connecting) points can be used jointly, linking the two associated meridians (external-internal) in such a way that, after assessing the state of a meridian's path, its Yuan point will be combined with the Luo point of its coupled meridian and vice versa; all this depending on the condition of the muscle fibres and on the path that wants to be treated for these. Generally, it is used to transfer energy from one meridian to the other and vice versa, depending on the condition presented by the patient.

The needles used for the treatments will be single-use needles of two different gauge sizes. One size or the other will be used depending on the area to be treated and the physical condition of the patient. The needles and gauge sizes used in the study are as follows:

Dong Bang siliconized needle 0.25 mm x 40 mm Dong Bang siliconized needle 0.20 mm x 30 mm

The therapist will assess the patient's condition according to traditional Chinese medicine and will look at the relationship between the patient's most affected areas and the paths of the acupuncture meridians. Subsequently, the combination of Yuan and Luo points to be treated will be determined. This procedure will be followed before every acupuncture session, in such a way that the combination of the points used will depend on the evolution of the symptoms.

Control group (C)

Sham acupuncture:

The course of action with the patient from the group that will use sham acupuncture will be the same as in the group that receives real treatment: patient in supine position, cleaning of the treated area, use of eye mask during the treatments and selection of points following the previously described Yuan and Luo points' criteria, based on traditional Chinese medicine.

The difference of sham acupuncture will lie on the way of performing the acupuncture technique. It will follow the validated technique of sham acupuncture with the Park device, without needle penetration in the patient's body.

The Park device for the performance of sham acupuncture consists of two plastic tubes, one sliding within the other, and inside which the needle created for the device slides. The longest tube is attached to a circular base, which has an adhesive surface that sticks to the skin so that the device and the needle cannot fall. Blunt ended needles will be used for this technique and thus the needle does not get to pass through the skin but produces a cutaneous stimulation similar to conventional acupuncture needles. These needles are supplied with the kit that contains the Park sham acupuncture device and are registered in the European Union as CE 0120.

Study variables

The main study variables are pain and quality of life.

Pain will be assessed using the Visual Analogue Scale (VAS). The VAS consisted of a 10 mm line with the endpoints 'no pain' and 'worst pain imaginable'.

The Fibromyalgia Impact Questionnaire (FIQ) will be used to analyse the quality of life. The FIQ is a multidimensional questionnaire designed specifically to assess the functional capacity of fibromyalgia patients. It is designed so that it can be self-administered by the patient. The values of the FIQ are between 0 and 100, 0 being the best state of health and 100 the worst. It takes five minutes to complete the FIQ. In this study, the Spanish version of the Revised Fibromyalgia Impact Questionnaire (FIQR) was used, which has proved its reliability and good construct validity.

The secondary variables are sleep quality and the subjective perception of participants regarding the effects of the treatment. The Medical Outcomes Study Sleep Scale (MOS-SS) will be used to assess the sleep quality. This specific questionnaire includes 12 items assessing data such as the quantity and quality of sleep. Items' responses were assigned scores using conventional scoring rules, with higher scores indicating a greater severity of sleep disturbance. The subjective perception of participants regarding the effects of the treatment will be assessed through the Patient Global Impression of Improvement Scale (PGI-I). The PGI-I consists of a single question in which patients are asked to classify the relief obtained with the treatment that they are following according to a seven-point scale from 'very much better to very much worse'. Only responses 'very much better' or 'much better' are associated with a successful treatment. All the other response options are defined as treatment failure.

These variables will be collected during the 8 weeks of the study, based on the individual interviews with the patients before each session and once the intervention is completed.

The interview with the patient will be conducted in the first session, when the physiotherapy clinical record will be created and the study tests will be taken for the first time. During the next 3 weeks, one weekly session of acupuncture will take place, thus adding up to 4 acupuncture sessions. Before the fourth study session, the tests will be taken again. Then, there will be another week of rest from interventions and, during the 6th week of the study, a new acupuncture intervention will be performed. One more week without intervention will then follow and the eighth week of the study will be only devoted to carrying out the tests in order to retrieve the survey data.

It is important to note that, in this last week of the study, a particular test will be conducted for the first time: the one related to the patient's impression of improvement with the treatment (PGI-I).

The data will be collected by researcher #2, blinded to the specific intervention group the subjects belong to.

Calculation of sample size

Acupuncture is considered to be effective in pain management if improvement according to the VAS scale is equal to or greater than 20%. On the basis of previous studies, it has been calculated that, in order to obtain an alpha error of 0.05 and a study power of 80%, a sample of 90 people is required (45 per group). Since a dropout of 10% is foreseen, this number has been extended to 100 (50 per group).

Statistical analysis

Demographic and basal variables will be defined using different measures. For a quantitative variable, the following will be used: mean, standard deviation and confidence interval at 95%. In addition to this, in case the variable did not have normal distribution, more robust descriptive statistics will be foreseen for the calculations, such as the median, the interquartile range and the minimum and maximum values. In the case of a qualitative variable, a frequency distribution will be drawn.

In order to assess potential changes in the instruments and scales used in the study over time, contrasts for dependent variables will be used, namely the ANOVA test for repeated measures or the Friedman test, depending on whether or not the distribution of the variable is normal. The Shapiro-Wilks test will be used for the normality test.

On the other hand, if differences existed among the different moments in which the instrument is evaluated, the ANOVA test for repeated measures will allow for the analysis of whether these differences are the same or different depending on the type of intervention performed.

Similarly, a variable that assesses changes in the main variables during the study will be created and a non-parametric contrast will be done in order to analyse whether such changes have been equal among the two groups. To finalise, a multivariate model will be applied in order to verify whether the intervention group has improved the parameters to be measured (linear or logistic regression depending on the dependent variable's nature). Such a model will be validated through the standard procedures.

Processing of data

In order to ensure a proper collection and processing of the data obtained, these will be managed by qualified staff from the same university and will be implemented by the clinical research coordinator.

Safety

Participants in the study will be controlled at all times against any adverse effects or complications, such as swelling, pain, hematomas in the needle insertion areas, discomfort, dizziness or heart palpitations after receiving the treatment. After every session and before starting the next one, questions will be asked to the participants and a visual inspection will be carried out in order to assess the potential undesirable effects of the last intervention.

Ethical principles

The Clinical Research Ethics Committee (CREC) of the Hospital Universitario Sant Joan de Reus has approved this protocol under approval reference number (15-07-30/7aclaproj1). The patients' data will be protected and will only be used for the purposes of this research.

ELIGIBILITY:
Inclusion Criteria:

* • Meeting the criteria set by the American College of Rheumatology for the diagnosis of chronic widespread pain.

  * Accepting to sign the informed consent of participation in the study.
  * Being older than 18 years.

Exclusion Criteria:

* Suffering from malignant diseases or active rheumatologic disorders (osteoporosis, rheumatoid arthritis, lupus erythematosus, etc.).

  * Suffering from coxarthrosis or severe gonarthrosis.
  * Having previously received acupuncture treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05-31 (Estimated); Study Completion 2017-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain will be assessed using the Visual Analogue Scale (VAS). | up to 8 weeks
  The VAS consisted of a 10 mm line with the endpoints 'no pain' and 'worst pain imaginable' .
The Fibromyalgia Impact Questionnaire (FIQ) will be used to analyze the quality of life. | up to 8 weeks

SECONDARY OUTCOMES:
The Medical Outcomes Study Sleep Scale (MOS-SS) will be used to assess the sleep quality. | up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Casado Borrull, Director, Principal Investigator
Locations (1):
- EUSESTE Escola Universitaria de la Salut i l'Esport Terres del'Ebre, Tortosa, Tarragona, Spain